CLINICAL TRIAL: NCT00976404
Title: Multicenter, Randomized, Non-comparative, Controlled Study of Therapeutic Intensification Plus Immunomodulation in HIV-infected Patients With Long-term Viral Suppression
Brief Title: Therapeutic Intensification Plus Immunomodulation to Decrease the HIV-1 Viral Reservoir
Acronym: EraMune02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert L. Murphy (Other)
Collaborators: Objectif Recherche Vaccins SIDA (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Robert L. Murphy, Professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EraMune02
Record Dates: First submitted 2009-09-09; First posted 2009-09-14 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infection
Keywords: HIV-1 infection; Treatment intensification; Immunomodulation; HIV-rAd5 vaccine
MeSH Terms: conditions — HIV Infections | interventions — DNA; Raltegravir Potassium; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc + raltegravir intensification (Active Comparator): ART Intensification (addition of raltegravir and maraviroc to suppressive ART for 56 weeks)
  Interventions: Drug: ART intensification (raltegravir); Drug: ART intensification (maraviroc)
- Maraviroc + raltegravir intens. plus DNA + HIV-rAd5 vaccine (Experimental): ART Intensification (addition of raltegravir and maraviroc for 56 weeks) PLUS immunomodulation therapy with DNA prime vaccine (Weeks 8,12,16) + HIV-recombinant Ad5-based vaccine (Week 32)
  Interventions: Biological: DNA + HIV-rAd5 vaccine; Drug: ART intensification (raltegravir); Drug: ART intensification (maraviroc)

INTERVENTIONS:
Biological: DNA + HIV-rAd5 vaccine — 4 mg subcutaneous injection at weeks 8 (DNA prime), 12 (DNA prime), 16 (DNA prime), and 32 (HIV-rAd5)
  Arms: Maraviroc + raltegravir intens. plus DNA + HIV-rAd5 vaccine
Drug: ART intensification (raltegravir) — raltegravir 400 mg PO BID for 56 weeks
  Other Names: Isentress
Drug: ART intensification (maraviroc) — maraviroc 150, 300, or 600 mg PO BID (depending on PK interactions with other medications) for 56 weeks
  Other Names: Selzentry; Celsentri

SUMMARY:
The objective of this study is to discover a new approach in which human immunodeficiency virus (HIV) can be eradicated from an infected individual by intensified antiretroviral treatment coupled with immunomodulation. The hypothesis is that eradication is possible only if very potent antiretroviral drugs are delivered in conjunction with an immunomodulatory agent that simultaneously attack the viral reservoirs.

DETAILED DESCRIPTION:
The objective of this study is to measure the impact of immunomodulation plus treatment intensification on the HIV reservoir in HIV-infected patients who have viral suppression on combination antiretroviral therapy. Treatment regimens first will be intensified by the addition of raltegravir and maraviroc for 8 week followed by immunomodulation with the NIH HIV-rAd5 vaccine plus DNA prime-boost for 24 weeks. The primary endpoint is measurement of change in peripheral cellular HIV DNA. A decrease of 0.5 log is considered significant. A secondary endpoints include change in HIV DNA in the rectal mucosa, immunologic changes in the peripheral blood and safety.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* At least 3 years of ART without interruption (less than one month cumulative)
* ART regimen unchanged in the 3 months prior to screening
* One HIV plasma viral load (RNA) documented at least 3 years prior to entry, and at least 2 HIV plasma viral load (RNA) documented per year thereafter
* HIV plasma viral load (RNA) ≤ 500 copies/mL at least 3 years prior to entry, and HIV plasma viral load < 500 copies/mL for >90% of the measures thereafter
* HIV plasma viral load (RNA) below the limit of detection for all values within the past year (one virologic blip allowed)
* HIV plasma viral load below the limit of detection within 60 days of entry
* CD4+ count ≥ 350 cells/mm3 within 60 days of entry
* Proviral DNA ≥10 and ≤1000 copies/106 PBMCs within 75 days of entry
* Adeno5 neutralizing antibody titers of 250 or less within 75 days of entry
* Hemoglobin ≥ 10 g/dL within 60 days of entry
* Platelets ≥ 100,000 per microliter within 60 days of entry
* Hepatic transaminases (ALT and AST) ≤ 2.5 x ULN within 60 days of entry
* Creatinine clearance > 50 mL/min by the Cockcroft-Gault equation within 60 days of entry

Exclusion Criteria:

* Sexually active men and women who will not practice at least one form of barrier birth control (male partner using condoms, female partner using condoms, other barrier contraception, etc)
* Pregnancy
* Inability or unwillingness to provide informed consent
* HBsAg positive
* HCV antibody positive or HCV RNA detectable
* Previous use of an integrase inhibitor (ie raltegravir) or a CCR5 inhibitor (ie maraviroc, vicriviroc). Use of raltegravir for non-treatment failure indications such as intensification or toxicity switches is allowed.
* Immunologic therapeutic intervention (e.g. IL-2) within the past year
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* Diagnosis of cancer within the last 5 years (except basal cell cutaneous cancers and cutaneous KS not requiring systemic therapy)
* Co-morbid condition with an expected survival of less than 12 months
* History of hypersensitivity to vaccination
* History of autoimmune disease, such as systemic lupus erythematosis (SLE) or Hashimoto's thyroiditis
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, MD, Study Chair — Northwestern University
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Cornell University, New York, New York

REFERENCES:
- [Derived] Achenbach CJ, Assoumou L, Deeks SG, Wilkin TJ, Berzins B, Casazza JP, Lambert-Niclot S, Koup RA, Costagliola D, Calvez V, Katlama C, Autran B, Murphy RL; EraMune 02 study team. Effect of therapeutic intensification followed by HIV DNA prime and rAd5 boost vaccination on HIV-specific immunity and HIV reservoir (EraMune 02): a multicentre randomised clinical trial. Lancet HIV. 2015 Mar;2(3):e82-91. doi: 10.1016/S2352-3018(15)00026-0. Epub 2015 Feb 17. PMID 26424549

RESULTS

PARTICIPANT FLOW:
Groups:
- ART Intensification: Maraviroc + Raltegravir: ART Intensification (addition of raltegravir and maraviroc) to suppressive ART for 56 weeks
- Maraviroc + Raltegravir Plus DNA + HIV-rAd5 Vaccine: ART Intensification (addition of raltegravir and maraviroc for 56 weeks) PLUS immunomodulation therapy with DNA prime vaccine (Weeks 8,12,16) + HIV-recombinant Ad5-based vaccine (Week 32)
Period: Overall Study
Arm/Group | ART Intensification: Maraviroc + Raltegravir | Maraviroc + Raltegravir Plus DNA + HIV-rAd5 Vaccine
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ART Intensification: Maraviroc +Raltegravir: ART Intensification (addition of raltegravir and maraviroc to suppressive ART for 56 weeks)
- Total: Total of all reporting groups
Arm/Group | ART Intensification: Maraviroc +Raltegravir | Maraviroc + Raltegravir Plus DNA + HIV-rAd5 Vaccine | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [46 to 55] | 50 [46 to 55] | 50 [46 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
CD4 cell count [Median (Inter-Quartile Range); unit: cells per mm^3] | 686 [501 to 880] | 563 [468 to 718] | 636 [485 to 791]
Time on antiretroviral treatment (ART) [Median (Inter-Quartile Range); unit: years] | 13 [8 to 19] | 13 [6 to 19] | 13 [8 to 19]
Adenovirus 5 antibody [Median (Inter-Quartile Range); unit: titer] — Serum Ad5 90% neutralization antibody titer
  titer | 18 [12 to 68] | 12 [12 to 38] | 12 [12 to 41]
HIV DNA [Median (Inter-Quartile Range); unit: copies per 10^6 PBMC] | 97 [47 to 352] | 228 [98 to 383] | 170 [60 to 361]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HIV DNA in PBMCs at Week 56
Time Frame: 56 weeks
Measure: Median (Inter-Quartile Range); unit: log^10 copies per 10^6 PBMCs
Arm/Group | ART Intensification: Maraviroc +Raltegravir | Maraviroc + Raltegravir Plus DNA + HIV-rAd5 Vaccine
Number analyzed (Participants) | 14 | 14
log^10 copies per 10^6 PBMCs | 0.00 [-0.29 to 0.16] | 0.04 [-0.11 to 0.19]

2. Secondary Outcome: Change From Baseline in HIV DNA in Rectal Tissue at Week 56
Time Frame: Week 56
Measure: Median (Inter-Quartile Range); unit: log^10 copies per 10^6 cells
Arm/Group | Maraviroc + Raltegravir Intensification | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine
Number analyzed (Participants) | 7 | 6
log^10 copies per 10^6 cells | 0.08 (0.27) [-0.06 to 0.22] | -0.02 (0.37) [-0.02 to 0.41]

3. Secondary Outcome: Change From Baseline in CD4+ T Cell Count at Week 56
Time Frame: Week 56
Measure: Median (Inter-Quartile Range); unit: cells per mm^3
Arm/Group | Maraviroc + Raltegravir Intensification | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine
Number analyzed (Participants) | 14 | 14
cells per mm^3 | -1 [-144 to 151] | 23 [-100 to 114]

4. Secondary Outcome: HIV Specific T-cell Response to Env
Description: HIV-specific immunity: Interferon gamma ELISpot response to Env (clades A) at week 36 (one month after rAd5 boosting)
Time Frame: 36 weeks
Measure: Median (Standard Deviation); unit: response per 10^6 PBMCs
Arm/Group | Maraviroc + Raltegravir Intensification | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine
Number analyzed (Participants) | 14 | 14
response per 10^6 PBMCs | 28 (50) | 86 (235)

5. Secondary Outcome: Serious Adverse Events Attributed to Study Treatments
Description: Grade 3 or 4 serious adverse events related to study treatments (raltegravir, maraviroc, or HIV-recombinant Ad5-based vaccine)
Time Frame: 56 weeks
Measure: Number; unit: serious adverse events
Arm/Group | Maraviroc + Raltegravir Intensification | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine
Number analyzed (Participants) | 14 | 14
serious adverse events | 1 | 3

ADVERSE EVENTS:
Time Frame: 56 weeks
Arm/Group | Maraviroc + Raltegravir Intensification | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc + Raltegravir Intensification (N=14) | Maraviroc + Raltegravir Intens. Plus DNA + HIV-rAd5 Vaccine (N=14)
creatine kinase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 4 creatine kinase
acute coronary syndrome (Cardiac disorders) | 0 | 1 (1) — Grade 3 left arm, neck and chest pain
Renal failure (Renal and urinary disorders) | 0 | 1 (1) — Grade 4 acute renal failure, Grade 4 creatinine
deep vein thrombosis (Vascular disorders) | 0 | 1 (1) — Grade 3 deep vein thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No